CLINICAL TRIAL: NCT01759771
Title: Vitamin D3 Supplementation for Low-Risk Prostate Cancer: A Randomized Trial
Acronym: VD3PCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-007-12S; Pro00019745 (Other: Medical University of South Carolina IRB)
Record Dates: First submitted 2012-12-27; First posted 2013-01-03 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Vitamin D3; Active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): 4,000 IU of VD3 for one year
  Interventions: Drug: Vitamin D3
- Arm 2 (Placebo Comparator): placebo for one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — 4,000 IU of VD3 for at least one year
  Arms: Arm 1
Drug: Placebo — Placebo for at least one year
  Arms: Arm 2

SUMMARY:
Vitamin D promotes the differentiation of prostate cancer cells and maintains the differentiated phenotype of prostate epithelial cells. The results of the investigators' clinical studies indicate that vitamin 1,25 dihydroxyvitamin D3 (VD3) supplementation results in a decrease of positive cancer cores at repeat biopsy in subjects with low-risk prostate cancer. The investigators hypothesize that Veterans who have early-stage prostate cancer and who take vitamin D3 at 4000 international units per day (intervention group) will show an improvement in the number of positive cores and in Gleason score at repeat biopsy, and a decreased likelihood of undergoing definitive treatment (prostatectomy or radiation therapy), compared to Veteran subjects taking placebo (control group).

DETAILED DESCRIPTION:
The central hypothesis of this grant application is that vitamin D3 (cholecalciferol) supplementation will benefit Veteran subjects diagnosed with early-stage, low-risk prostate cancer, who elect to have their disease monitored through active surveillance. Specifically, the investigators hypothesize that Veterans who take vitamin D3 at a daily dose of 4000 international units (IU) for a minimum of one year (intervention group) will show an improvement in the number of positive cores and in Gleason score at repeat biopsy, and a decreased likelihood of undergoing additional treatment (hormone therapy, prostatectomy or radiation therapy), compared to Veterans taking placebo (control group).

To test this hypothesis, the investigators propose the following Specific Aims:

1. To determine whether vitamin D3 (4,000 IU per day FOR AT LEAST ONE YEAR) will result in a significant improvement of the pathology status at repeat biopsy in Veteran subjects taking vitamin D3, compared to Veteran subjects taking placebo. This hypothesis will be tested through a randomized clinical trial, which will enroll 136 Veteran subjects (68 participants per arm), diagnosed with early-stage prostate cancer (Gleason score 6, PSA 10, clinical stage T1C or T2a). The pathology status will be measured by the change in Gleason score and the number of positive cores in prostate needle biopsy specimens between baseline and the end of the study. Pre- and post-study biopsies will be performed as part of the standard medical care for diagnosis and active surveillance.
2. To determine whether vitamin D3 supplementation, compared to placebo, will result in a significant decrease in the number of Veteran subjects who will undergo additional treatment (hormone therapy, prostatectomy or radiation therapy), following the outcome of repeat biopsy.
3. To analyze changes in the serum levels of cholecalciferol, 25(OH)D, 1,25(OH)2D, and prostate-specific antigen (PSA) at baseline and at the end of the study, and to estimate the associations between changes in these measures and pathology outcomes (Gleason score and number of positive cores).
4. To compare the expression of molecular biomarkers, which are prognostically relevant to prostate cancer progression, in pre- and post- treatment biopsy tissue specimens. Paraffin-embedded sections will be processed to assess by immunohistochemical techniques the expression of the following biomarkers: Vitamin D Receptor (VDR), P21, Tumor Growth Factor (TGF ), Cyclooxygenase 2 (COX-2), and NF B. All of these protein products impact growth control and chronic inflammation in prostate cancer progression and are specifically affected by Vitamin D status.

Implementation of the proposed studies would demonstrate that Vitamin D3 supplementation provides a welcome addition to active surveillance, since patients who respond to Vitamin D3 supplementation (as indicated by a decrease in score or number of positive cores at repeat biopsy) can safely continue active surveillance and would not need definitive treatment. In turn, this would result in a decreased likelihood of overtreatment. On the other hand, subjects who progress after Vitamin D3 supplementation, as indicated by an increase in Gleason score or number of positive cores at repeat biopsy, may have more aggressive disease and may need to consider definitive treatment. Therefore, both groups of patients (responders as well as non-responders) would benefit from Vitamin D3 supplementation, an intervention strategy that is extremely cost-effective and easy to implement.

ELIGIBILITY:
Inclusion Criteria:

* Male 19 - 90 years old - Low-grade prostate cancer
* Clinical Stage T1C or T2a
* Serum PSA < 10.0 ng/ml
* Gleason Score < or = to 6 (either architectural pattern < or = to 3)
* Decision to monitor prostate cancer in Active Surveillance
* Serum creatinine < 2.0 mg/dL
* Serum phosphorus > 2.3 and < 4.8 mg/dL
* Serum calcium > 8.5 and < 10.5 mg/dL
* Must be capable of giving consent to participate in the study

Exclusion Criteria:

* Any concurrent malignancy, except non-melanoma skin cancer
* History of sarcoidosis
* History of Primary Hyperparathyroidism
* History of hypercalcemia
* Vitamin D supplementation > 2,000 IU daily
* Lithium medication

Ages: 19 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Diagnosis of Early-stage Prostate Cancer
Enrollment: 130 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Gattoni-Celli, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 58 | 56
Completed | 57 | 55
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 22 | 67
  >=65 years | 13 | 34 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 56 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 20 | 42
  White | 36 | 36 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 56 | 114
Prostate specific antigen [Mean (Full Range); unit: ng/ml] | 5.64 [1.13 to 9.8] | 6.03 [0.46 to 13.4] | 5.83 [0.46 to 13.4]
Gleason Score [Mean (Full Range); unit: units on a scale] — Gleason score goes from 6-10, with 6 being the lowest and 10 being the highest. Lower portends a better prognosis and higher portends a worse prognosis. The Gleason score is determined by the pathologist viewing the histopathology of the biopsy who assesses the architectural pattern of the cancer. This is an agreed upon scale to communicate what is often described as grade in other, non-prostate, cancers.
  units on a scale | 6 [6 to 6] | 6 [6 to 6] | 6 [6 to 6]
Parathyroid hormone [Mean (Full Range); unit: pg/ml] | 57.5 [17 to 129] | 56.03 [16 to 124] | 56.8 [16 to 129]
25(OH)D3 [Mean (Full Range); unit: ng/ml] | 29.37 [11.8 to 55.5] | 26.98 [7 to 53.8] | 28.20 [7 to 55.5]
Number of positive cores [Mean (Full Range); unit: positive cores] — The standard of care is taking 12 biopsy cares. A commonly reported statistic includes how many of these 12 cores are positive. As such, this would be a unit of measure anywhere from 0-12 cores positive. A higher number of positive cores is prognostically more concerning than a lower number of positive cores. For patients on active surveillance, an increase in the number of positive cores will often prompt treatment rather than continuing with observation.
  positive cores | 2.43 [1 to 8] | 1.95 [1 to 5] | 2.23 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Pathology Status
Description: pathology status will be measured by the number of positive cores in prostate needle biopsy specimens between baseline and the repeat standard of care prostate biopsy at the end of the study.
Time Frame: one year
Measure: Mean (Full Range); unit: number of positive cores
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 58 | 56
number of positive cores | 2.37 [0 to 11] | 1.73 [0 to 7]

2. Secondary Outcome: Number of Veteran Subjects Who Will Undergo Additional Treatment
Description: To determine whether vitamin D3 supplementation, compared to placebo, will result in a significant decrease in the number of Veteran subjects who will undergo additional treatment (prostatectomy or radiation therapy), following the outcome of repeat biopsy.
Time Frame: 2 years
Population: Analysis of population receiving vitamin D supplementation vs placebo and assessing those who move on to treatment of prostate cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 58 | 56
Participants | 15 | 18

3. Secondary Outcome: PSA and Serum Vitamin D
Description: To analyze changes in the serum levels of cholecalciferol, 25(OH)D, 1,25(OH)2D, and prostate-specific antigen (PSA) at baseline and at the end of the study.
Time Frame: One year
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 58 | 56
ng/ml
  24(OH)D3 | 48.68 [26.5 to 100.7] | 26.98 [7 to 53.8]
  PSA | 6.084 [1.02 to 12.02] | 6.25 [0.88 to 14.02]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over the period of the study which was 12 months.
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 0/58 | 0/56

LIMITATIONS AND CAVEATS:
The study is limited by the potential challenges associated with needle biopsy as opposed to full pathologic specimens.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-08-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT01759771/Prot_SAP_000.pdf